CLINICAL TRIAL: NCT04404400
Title: Hydrocortisone and Fludrocortisone for Critical Illness-related Corticosteroid Insufficiency
Acronym: HORNbILL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP200018; 2020-003942-35 (EudraCT Number)
Record Dates: First submitted 2020-05-19; First posted 2020-05-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Critical Illness Related Corticosteroids Insufficiency
Keywords: critical illness related corticosteroids insufficiency; hydrocortisone; fludrocortisone; ICU; survival

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): For CIRCI patients: hydrocortisone + fludrocortisone therapy.
  Interventions: Drug: Investigational products administration
- Placebo (Placebo Comparator): For CIRCI patients: hydrocortisone placebo + fludrocortisone placebo
  Interventions: Drug: Placebo administration

INTERVENTIONS:
Drug: Investigational products administration — Investigational products include:
  * Hydrocortisone hemisuccinate 50 mg: one intravenous injection every 6 hours, and
  * 9 alpha fludrocortisone 50 μg: one tablet per day via a nasogastric tube.
  All treatments will be stopped after 7 days or until the patient has left the intensive care unit (whichever occurs first) without tapering off.
  Arms: Active
Drug: Placebo administration — Placebos for hydrocortisone and for fludrocortisone, administered in same manner as the active drugs in the interventional arm, for 7 days.
  Arms: Placebo

SUMMARY:
The study aims at assessing the efficacy and the safety of hydrocortisone combined with fludrocortisone compared to placebo in ICU adults with critical illness related corticosteroid insufficiency.

DETAILED DESCRIPTION:
The hypothalamic-pituitary-adrenal axis together with the noradrenergic/vasopressinergic system are the main systems of host response to stress. In 2008 the scientific community described a syndrome called critical illness related corticosteroids insufficiency (CIRCI) in which body homeostasis is lost owing to insufficient cortisol production or bioactivity in tissues. Recent updates of international guidelines have spelled out the pathophysiology, diagnosis and management of CIRCI. The prevalence of CIRCI varies according to case mix and severity of illness. The combination of hydrocortisone and fludrocortisone improved outcomes in septic shock, a condition often complicated with CIRCI. However, there is insufficient evidence on the efficacy of corticosteroids in patients with CIRCI and without septic shock. The hypothesis of the study is that the hydrocortisone-fludrocortisone association will improve ventilation and vasopressor free survival in ICU patients with Critical illness related Corticosteroid Insufficiency.

Patients with a SOFA score ≥ 4 will be screened for CIRCI. Patients suffering from CIRCI will be randomized to receive hydrocortisone and fludrocortisone or their placebo. Patients without CIRCI will receive standard of care and will be followed up during 90 days (cohort-observational study).

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥ 18 years);
* Hospitalized in an intensive care unit;
* SOFA score ≥ 4, for at least 6 consecutive hours;
* Informed written consent from patient or from legally authorized next of kin, or emergency deferred consent;
* Affiliation to a social security system or to a universal health coverage (Couverture Maladie Universelle, CMU).

Exclusion Criteria:

* Any suspected or proven acute adrenal insufficiency (As defined in international guidelines; basal cortisol < 5 μg/dL or peak (60) cortisol <18 μg/dL)
* Expected death or withdrawal of life-sustaining treatments within 48 hours
* Known chronic adrenal insufficiency
* Concomitant treatment that inhibits cortisol production
* Septic shock (Singer Jama 2016)
* Active tuberculosis or fungal infection
* Active viral hepatitis or active infection with herpes viruses
* Hypersensitivity or contraindication to hydrocortisone, fludrocortisone or Synacthène® or any of their excipients ( SmPC)
* Patient needing either anti-inflammatory corticosteroids or substitutive hydrocortisone for any reason (Such as those suffering from COVID-19 pneumonia requiring oxygen therapy).
* Current treatment by more than 15 mg/d of prednisone (or equivalent) for more than 30 days
* Diabetic ketoacidosis or hyperglycemic hyperosmolar syndrome
* Pregnant or breastfeeding woman
* Moribund patient
* Previously enrolled in this study
* Participation to another interventional study that focuses on CIRCI and/or corticoid drugs and/or that addresses a similar primary endpoint as Hornbill ( ventilator- and vasopressor-free survival )
* Patient under guardianship or tutorship

Note: Included patients for whom acute adrenal insufficiency would be detected in the Synacthen ® test performed as part of the research for the diagnosis of CIRCI will not be randomized since they should be treated by corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1092 (Estimated)
Dates: Start 2022-02-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
number of ventilator- and vasopressor-free days | at day 30
  number of ventilator- and vasopressor-free days within 30 days (deaths assigned zero days) after randomisation.

SECONDARY OUTCOMES:
Mortality rates | at day 30, 90 and 180
  Mortality rates at ICU and hospital discharge and at day 30, 90 and 180 after randomization
Number of days alive without vasopressors | at day 30
  Number of days alive without vasopressors on day 30 after randomization.
Number of days alive free of mechanical ventilation | at day 30
  Number of days alive free of mechanical ventilation on day 30 after randomization.
Number of days alive with SOFA < 4 | daily un to 30 days
  Number of days alive with SOFA < 4 in the 30 days after randomization
Withhold and/or withdraw proportion | up to 3 months
  Proportion of patients with a decision to withhold and/or withdraw active treatments.
ICU duration | up to 3 months
  Duration of stay (unit: day and minutes) at ICU.
duration of hospitalization of stay | daily up to 30 days
  Duration of hospitalization of stay.
Rate of re-admission to the ICU | daily up to 30 days
  Rate of re-admission to the ICU during the 30 days after randomization.
Safety endpoints - serious adverse events associated with corticosteroids | daily up to 30 days
  - Proportion of patients affected by any serious adverse events associated with corticosteroids, among the following: hospital-acquired infections, hyperglycemia, hypernatremia, neurological disorders (coma, stroke or muscle weakness) during the 30 days after randomization.
Safety endpoints - hospital-acquired infections proportion | daily up to 30 days
  - Proportion of patients affected by hospital-acquired infections;
Safety endpoints - hyperglycemia | daily up to 30 days
  - Number of episodes of hyperglycemia during ICU stay or up to day 30, whichever occurs first;
Safety endpoints - hypernatremia | daily up to 30 days
  - Number of episodes of hypernatremia during ICU stay or up to day 30, whichever occurs first;
Safety endpoints - Gastroduodenal bleeding | daily up to 30 days
  - Gastroduodenal bleeding requiring transfusion or hemostatic treatment during ICU stay or up to day 30, whichever occurs first;
Safety endpoints - corticosteroids administration requiring | daily up to 30 days
  - Number of patients requiring the administration corticosteroids following the end of the administration of the experimental treatment.
Rate of ventilation and vasopressors free survival at day 90 | at day 90
  Secondary endpoint concerning screened but non-randomised patients:
  Rate of ventilation and vasopressors free survival at day 90 in subjects devoid of CIRCI
Renal replacement therapy (RRT)-free days | up to day 30
  Renal replacement therapy (RRT)-free days up to Day 30 after randomisation (excluding patients on RRT for chronic renal failure at time of randomisation)
response to glucocorticoids | up to 3 months
  Score of cutaneous vasoconstrictor response to glucocorticoids
Change in quality of life | up to Day 30 and 90
  Change in utility, based on the EuroQol group's 5-dimension 5-level (EQ-5D-5L) questionnaire, up to Day 30 and 90 after randomisation
Rate of ventilation | at day 30
  Endpoint concerning non-randomised patients:
  Rate of ventilation at day 30 post SYNACTHENE® test
Vasopressors free days | at day 30
  Endpoint concerning non-randomised patients:
  Vasopressors free days at day 30 post SYNACTHENE® test

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas HEMING, MD, PhD, Principal Investigator — General Intensive care Unit, Raymond Poincaré Hospital, APHP; Djillali ANNANE, MD, PhD, Study Director — General Intensive care Unit, Raymond Poincaré Hospital, APHP
Locations (1):
- General Intensive care Unit, Raymond Poincaré Hospital, APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Annane D, Pastores SM, Rochwerg B, Arlt W, Balk RA, Beishuizen A, Briegel J, Carcillo J, Christ-Crain M, Cooper MS, Marik PE, Umberto Meduri G, Olsen KM, Rodgers S, Russell JA, Van den Berghe G. Guidelines for the diagnosis and management of critical illness-related corticosteroid insufficiency (CIRCI) in critically ill patients (Part I): Society of Critical Care Medicine (SCCM) and European Society of Intensive Care Medicine (ESICM) 2017. Intensive Care Med. 2017 Dec;43(12):1751-1763. doi: 10.1007/s00134-017-4919-5. Epub 2017 Sep 21. PMID 28940011
- [Background] Annane D, Renault A, Brun-Buisson C, Megarbane B, Quenot JP, Siami S, Cariou A, Forceville X, Schwebel C, Martin C, Timsit JF, Misset B, Ali Benali M, Colin G, Souweine B, Asehnoune K, Mercier E, Chimot L, Charpentier C, Francois B, Boulain T, Petitpas F, Constantin JM, Dhonneur G, Baudin F, Combes A, Bohe J, Loriferne JF, Amathieu R, Cook F, Slama M, Leroy O, Capellier G, Dargent A, Hissem T, Maxime V, Bellissant E; CRICS-TRIGGERSEP Network. Hydrocortisone plus Fludrocortisone for Adults with Septic Shock. N Engl J Med. 2018 Mar 1;378(9):809-818. doi: 10.1056/NEJMoa1705716. PMID 29490185